CLINICAL TRIAL: NCT06352749
Title: Face-to-face vs Online Physical Exercise in Seniors Living in Nursing Homes: Randomized Controlled Trial on Its Effects on Health and Quality of Life
Brief Title: Face-to-face vs Online Physical Exercise in Seniors Living in Nursing Homes (ExerMOT-NH)
Acronym: ExerMOT-NH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Collaborators: Fundación Miranda (Unknown); Residencia Albiz Santiago Llanos (Unknown); Aspaldiko (Unknown); Residencia Nuestra Señora de Begoña, Santurtzi (Unknown)
Responsible Party: Principal Investigator, Jon Irazusta, Professor, University of the Basque Country (UPV/EHU)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BasqueCU2024
Record Dates: First submitted 2024-03-17; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Physical Function; Cognitive Decline; Psychological Well-Being
Keywords: physical exercise; online; nursing homes; older adults
MeSH Terms: conditions — Cognitive Dysfunction; Psychological Well-Being; Motor Activity

STUDY DESIGN:
Intervention Model Description: Each group will be assigned to control, online intervention or face-to-face intervention
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigators in charge of doing the statistical analysis and assessing the outcome measures will be blinded to group allocation. Due to the characteristics of the study, blinding the participants and the care provider (i.e., the professional conducting the exercise sessions) to the group allocation is not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Sham Comparator): Participants will receive advice to be physically active and to reduce their sedentary behavior
  Interventions: Behavioral: Advice to increase physical activity and reduce sedentary behavior
- Online exercise (Experimental): Participants will receive general recommendations for maintaining physically active and reducing sedentary behaviors. This will be done verbally and through written material. In addition, participants will take part in a 6-month multicomponent physical exercise program consisting of 2 online weekly multicomponent sessions.
  Interventions: Behavioral: Advice to increase physical activity and reduce sedentary behavior; Behavioral: Online Physical Exercise
- Face-to-face exercise (Active Comparator): Participants will receive general recommendations for maintaining physically active and reducing sedentary behaviors. This will be done verbally and through written material. In addition, participants will take part in a 6-month multicomponent physical exercise program consisting of 2 face-to-face weekly multicomponent sessions.
  Interventions: Behavioral: Advice to increase physical activity and reduce sedentary behavior; Behavioral: Face-to-Face Exercise

INTERVENTIONS:
Behavioral: Advice to increase physical activity and reduce sedentary behavior — After the baseline assessments, all participants will receive individualized counseling for following physically active lifestyle and reducing sedentary behaviors. Participants will be encouraged to increase the physical activity time and intensity, and to hourly break the sedentary time while at home. The recommendations will be transmitted verbally and through written material.
Behavioral: Online Physical Exercise — This intervention will entail:
  Strength training of upper and lower limbs. Familiarization phase will include 2-3 exercises of 1-2 series and 8-12 repetitions per session. During the acquisition phase, 2-3 exercises of 2-3 series and 8-12 repetitions at a higher velocity. The resting time between sets will be of 1-3 minutes.
  Balance exercises will include proprioception, agility and weight transfer exercises. Difficulty will progressively increase by reducing the base of support, by including multidirectional displacements, walking on tiptoe or heels, body-weight transfer, dynamic exercises modifying the centre of gravity, and stressing postural muscles and by sensorial reductions.
  Flexibility exercises: Static stretching maintained during 20-30s carried out at the end of each session.
  All the sessions will be supervised online by trained physiotherapists or sports physiologists.
  Arms: Online exercise
Behavioral: Face-to-Face Exercise — This intervention will entail:
  Strength training of upper and lower limbs. Familiarization phase will include 2-3 exercises of 1-2 series and 8-12 repetitions per session. During the acquisition phase, 2-3 exercises of 2-3 series and 8-12 repetitions at a higher velocity. The resting time between sets will be of 1-3 minutes.
  Balance exercises will include proprioception, agility and weight transfer exercises. Difficulty will progressively increase by reducing the base of support, by including multidirectional displacements, walking on tiptoe or heels, body-weight transfer, dynamic exercises modifying the centre of gravity, and stressing postural muscles and by sensorial reductions.
  Flexibility exercises: Static stretching maintained during 20-30s carried out at the end of each session.
  All the sessions will be supervised face-to-face by trained physiotherapists or sports physiologists.
  Arms: Face-to-face exercise

SUMMARY:
The benefits of multicomponent physical exercise (MPE) in the mental and physical health of older adults are widely accepted. However, during Covid19 pandemic, some face-to-face programs for physical exercise were canceled. The situation was particularly complex in nursing homes (NHs) because residents were often confined to their floors and many leisure activities were canceled. Online physical exercise sessions increased their popularity during the pandemic. However, there is no evidence that online physical exercise sessions are an effective alternative to face-to-face sessions for older people living in NHs. The current project aims to assess a synchronous online MPE program's feasibility, acceptability, and effects. With this aim, first a synchronous online MPE intervention was designed and then a multicenter randomized controlled trial with 3 branches was developed: face-to-face MPE, online MPE and control. Participants in the control group will receive advice to maintain physical activity and reduce sedentary behavior. Additionally, those in the intervention groups will also participate in 24-week individualized and progressive MPE programs performed at moderate intensity that will be focused on strength, balance, and endurance. MPE will be performed through supervised sessions (2 per week). One of the intervention groups will be supervised face-to-face whereas the other will be supervised synchronously online. Study assessments will be conducted at baseline, at the end of the 24-week intervention, and after 24-week follow-up. The primary outcomes of the study will be changes in mental and physical health. Secondary outcomes will include other parameters of mental and physical health, together with physical activity, frailty, quality of life, and biological markers. The dropout rate, the adherence, the injuries and other adverse events suffered by the participants, and technical incidences produced in the online modality will be recorded. A mixed-model ANCOVA will be performed to compare the data between intervention and control groups, considering as co-variables baseline measurements. The statistical analysis will be performed on the whole sample and separated for sex/gender. The study received ethical approval (M10_2022_405_IRAZUSTA ASTIAZARAN). The results of this project will be transferred to institutions and entities involved in managing NHs to increase the opportunities for the residents to remain physically active.

ELIGIBILITY:
Inclusion Criteria:

* Older than 65 years
* A score equal to or higher than 15 out of 35 in the MEC-35 (Miniexamen Cognoscitivo) cognitive test
* A score equal to or higher than 50 out of 100 in the Barthel Index
* Able to stand-up and walk for 10 meters

Exclusion Criteria:

* Unstable Clinical Situation
* When the potential harms outweigh the benefits, according to the judgment of the healthcare personnel at the NHs

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Trail Making Test (TMT) | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  The TMT is a valid and widely used test to assess executive functioning. The TMT consists of two parts, part A and part B. Part A is based on number sequencing and assesses visual-perceptual abilities and participants have to draw lines to link numbers from 1 to 25 in ascending order. Part B focus on number and letter switching evaluates cognitive flexibility and consists of drawing a line to link the numbers and the letters alternatively following in ascending order (e.g. 1-A-2-B-3-C). The completion time will be registered in seconds. Lower duration indicates better performance
Spanish Version of the Yesavage Depression Scale | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  The Yesavage Depression Scale, also known as the Geriatric Depression Scale (GDS), is a widely used self-report questionnaire designed to detect symptoms of depression in older adults. it consists 15 simple yes/no questions focusing on mood, cognition, and behavior. The scale helps assess the severity of depressive symptoms and can aid in determining the need for further evaluation or intervention. The scores range from 0 to 15. Higher values indicate more depressive symptoms.
30-seconds Chair Sit to Stand test | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  A test to measure muscle function of the lower limbs. Starting in a seated position, participants will be instructed to perform as many full sit-to-stand cycles as they could in a 30-second timeframe with the number of cycles considered the score for this test. Higher scores indicate better performance.

SECONDARY OUTCOMES:
MoCA (Montreal Cognitive Assessment) | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  MoCA test will be used to evaluate the cognitive function of participants. The MoCA was designed as a rapid screening instrument for mild cognitive dysfunction (63). It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. Time to administer the MoCA is approximately 10 minutes. The total possible score ranged from 0 to 30. Higher scores indicate better performance.
Wechsler Adult Intelligence Scale III (WAIS-III) | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  The WAIS-III is a test battery that has long been the gold standard for the evaluation of cognitive abilities (69). Specifically, we only use the digit span to evaluate working memory (70). Participants will be asked to recall a list of numbers in the order that they will be given (forward or backwards). The test is finished when for the same item the participant fails two attempts. A total number of correct answers will be registered for each condition. Higher values indicate better performance.
EuroQol-5 dimensions (EQ-5D-5L) | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  European Quality of Life-5 Dimensions (EQ-5D) questionnaire. Participants will self-rate their health on a vertical visual analogue scale (score range: 0-100), where the endpoints are labeled 'The worst health you can imagine' and 'The best health you can imagine'. Higher values indicate better quality of life.
The Spanish adaptation of the Basic Psychological Needs in Exercise Scale (BPNES) (Moreno et al., 2008) | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  The BPNES will be used to evaluate the satisfaction of the needs perceived by the participants (73). This questionnaire includes 12 items distributed in three dimensions (autonomy, competence and the other four items measure the relationship). The score ranges from 12 to 60. Higher values indicates a greater fulfillment of basic needs in physical exercise.
Zung's Anxiety Self-Assessment Scale (Hernández-Pozo, et al., 2008) | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  The Zung Anxiety Scale is a self-report questionnaire to measure the severity of anxiety symptoms in individuals. It consists of 20 questions related to various aspects of anxiety, such as physical symptoms, cognitive aspects, and emotional manifestations. Respondents rate each item based on how frequently they experience each symptom. The scale provides a quantitative assessment of anxiety levels, helping professionals to identify individuals experiencing significant anxiety symptoms and determine appropriate interventions.
Satisfaction with Life Scale | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  It is a 5-question scale with Likert-type answers of 5 categories that examines de global grade of satisfaction with life. Possible answers go from absolutely untrue (1) to absolutely true (5). A score of 5 to 25 points can be obtained. Higher values indicate better satisfaction with life. The score ranges from 5 to 35. Higher values indicate greater satisfaction.
Short Physical Performance Battery (SPPB) | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  The SPPB consists of three tasks that evaluate the lower extremities' function: balance, walking speed and sit-to-stand 5 times from a chair. In each task 0 to 4 points can be scored, to obtain a total score between 0 and 12 points. Higher values indicate better function.
The Biceps Curl Test | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  This requires people to repeatedly lift a 5 lb (2.27 kg) weight (for women) or an 8 lb (3.63 kg) weight (for men) for 30 seconds. The number of lifts is recorded. This reflects upper body strength. Higher values indicate better performance.
The 2-minute Walk Test (2-MWT) | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  2-MWT is an adaptation of 6-MWT. The test measured distance in meters walked in 2 minutes and reflects aerobic endurance. The original version of the Senior Fitness Test required people to walk on a rectangular course but more recent versions use a straight line. Higher values indicate better performance.
The 8 Feet Up-and-Go test | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  The test measures the time the subject needs to stand from a chair, walk 8 feet (2,5 meters), turn around, get back to the chair, and sit. The longer the time to complete the test, the worse the performance. Leaning on the thighs or the chair is allowed to stand. Lower time indicates better performance.
Handgrip strength test | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  The grip strength of each hand will be measured with a manual dynamometer. This variable is related to the general strength of the subject, where higher values indicate greater strength
Serum Brain Derived Neurotrophic Factor (BDNF) | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning after an overnight fast and at least 24 h after the last exercise session. After collection, tubes will be centrifuged at 5000 rpm for 10 min. Serum obtained for each participant will be stored in aliquots at -80 °C until analysis. Serum BDNF (ng/mL) will be quantified using a sandwich enzyme-linked immunosorbent assay (ELISA). Human BDNF Quantikine Immunoassay (R
  &D Systems, Minneapolis, MN) will be performed according to the manufacturer's instructions. Results will be reported as ng/mL.
Serum Klotho | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. Following collection, the tubes will be centrifuged at 5000×g for 10 min. The serum obtained from each participant will be stored in aliquots at - 80 °C for further analysis. A commercial enzyme-linked immunosorbent assay (ELISA) will be performed to measure klotho serum concentration according to the manufacturer's protocol (Human soluble α-Klotho Assay Kit JP27998, Immuno-Biological Laboratories Co., Ltd., Gunma, Japan). The quantification will be performed spectrophotometrically using a FLUOstar OPTIMA Microplate Reader (ThermoFisher Scientific, Waltham, MA, USA) and Optima Control software version 2.20. Results will be reported as ng/mL.
Serum Glucose | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The glucose concentration (mg/dL) will be measured in blood serum using routine clinical techniques.
Serum Urea | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The urea concentration (mg/dl) will be measured in blood serum using routine clinical techniques.
Serum Creatinine | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The concentration (mg/dL) will be measured in blood serum using routine clinical techniques.
Serum Uric Acid | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The uric acid concentration (mg/dL) will be measured in blood serum using routine
Serum Cholesterol | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The cholesterol concentration (mg/dL) will be measured in blood serum using routine clinical techniques.
Serum Triglycerides | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The triglyceride concentration (mg/dL) will be measured in blood serum using routine clinical techniques.
Serum HDL-Cholesterol | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The HDL-Cholesterol concentration (mg/dL) will be measured in blood serum using routine clinical techniques.
Serum LDL-Cholesterol | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The LDL-Cholesterol concentration (mg/dL) will be measured in blood serum using routine clinical techniques.
Serum Glutamate Pyruvate Transaminase | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. Serum glutamate pyruvate transaminase activity will be measured in blood serum using routine clinical techniques.
Serum Glutamate Oxaloacetate Transaminase | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The glutamate oxaloacetate transaminase activity will be measured in blood serum using routine clinical techniques.
Serum gamma glutamyl transferase | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The gamma glutamyl transferase activity will be measured in blood serum using routine clinical techniques.
Serum Alkaline Phosphatase | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The alkaline phosphatase activity will be measured in blood serum using routine clinical techniques.
Serum Creatin Kinase | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The creatin kinase activity will be measured in blood serum using routine clinical techniques.
Serum Lactate Dehydrogenase | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The lactate dehydrogenase activity will be measured in blood serum using routine clinical techniques.
Serum Bilirubin | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The bilirubin concentration (mg/dL) will be measured in blood serum using routine clinical techniques.
Serum Sodium | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The sodium concentration (mEq/L) will be measured in blood serum using routine clinical techniques.
Serum Potassium | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The potassium concentration (mEq/L) will be measured in blood serum using routine clinical techniques.
Serum Chloride | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The chloride concentration (mEq/L) will be measured in blood serum using routine clinical techniques.
Serum C Reactive Protein | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The C reactive protein concentration (mg/dL) will be measured in blood serum using routine clinical techniques.
Serum Albumin | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The albumin concentration (g/dL) will be measured in blood serum using routine clinical techniques
Serum Total Protein | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The total protein concentration (g/L) will be measured in blood serum using routine clinical techniques
Serum Calcium | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The calcium concentration (mg/dL) will be measured in blood serum using routine clinical techniques
Serum Phosphorus | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The phosphorus concentration (mg/dL) will be measured in blood serum using routine clinical techniques
Serum D Vitamin | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The D vitamin concentration (ng/dL) will be measured in blood serum using routine clinical techniques
Erythrocyte count | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The number of erythrocytes will be measured in blood using routine clinical techniques
Hemoglobin | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The hemoglobin concentration will be measured in blood using routine clinical techniques
Hematocrit | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The hematocrit will be calculated in blood using routine clinical techniques
Mean Corpuscular Volume (MCV) | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The mean corpuscular volume will be measured in blood using routine clinical techniques
Mean Corpuscular Hemoglobin (MCH) | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Baseline blood samples will be collected in the morning following an overnight fast. The mean corpuscular hemoglobin will be measured in blood using routine clinical techniques.
Mean Corpuscular Hemoglobin Concentration (MCHC) | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The mean corpuscular hemoglobin concentration will be measured in blood using routine clinical techniques
Red Cell Distribution Width (RDW) | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The red cell distribution width will be measured in blood using routine clinical techniques
Leucocyte Count | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The number of leucocytes will be measured in blood using routine clinical techniques
Neutrophil Count and Percentage | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The number of neutrophils will be measured in blood using routine clinical techniques. The percentage of neutrophils in the total white blood cell count will be calculated.
Lymphocyte Count and Percentage | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The number of lymphocytes will be measured in blood using routine clinical techniques. The percentage of lymphocytes in the total white blood cell count will be calculated.
Monocyte Count and Percentage | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The number of monocytes will be measured in blood using routine clinical techniques. The percentage of monocytes in the total white blood cell count will be calculated
Eosinophil Count and Percentage | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The number of eosinophils will be measured in blood using routine clinical techniques. The percentage of eosinophils in the total white blood cell count will be calculated
Basophil Count and Percentage | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The number of basophils will be measured in blood using routine clinical techniques. The percentage of basophils in the total white blood cell count will be calculated
Platelet Count | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The number of platelets will be measured in blood using routine clinical techniques.
Platelet Mean Volumen | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Blood samples will be collected in the morning following an overnight fast. The mean volume of platelets will be measured in blood using routine clinical techniques.
Physical activity, sedentary lifestyle and sleep will be evaluate using accelerometry | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Physical activity level was recorded with an accelerometer (Actigraph GT3X model; Actigraph LLC, Pensacola, FL, USA) that participants wore on the wrist with a belt for 7 days. Participants did not receive additional instructions to walk during the assessment period. The accelerometer was set to record the number of steps taken per day. Active-period intensities were classified as light, moderate, or vigorous, and were measured in minutes per day at each intensity. Sedentary time, bouts and breaks will be also recorded.
Fried's frailty phenotype score | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  Frailty will be analyzed with the 5 criteria suggested by Fried: unintentional weight loss, weakness or poor handgrip strength, self-reported exhaustion, slow walking speed, and low physical activity. The presence of each criterion will be scored with one point, the total score ranging between 0-5 points. A higher score indicates higher frailty.
Frail-NH frailty scale | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  It consist of 6 items Fatigue, resistance, ambulation, nutritional approach and help with dressing. Each item could receive a score from 0 to 2 and total score ranges from 0 to 13. An score < 6 is defined as non-frail; 6-7 as prefrail and > 7 as frail.
The Pittsburgh Sleep Quality Index | At baseline, after 24 weeks of intervention and after 24 weeks follow-up
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score. The Score ranges from 0 to 21. Higher values indicate worse sleep.
Attendance rate | During 24 weeks of intervention
  Attendance rate to face-to-face sessions will be calculated as the percentage of sessions attended out of the actual number of sessions offered. Reasons for non-attendance will be also provided
Dose modification | During 24 weeks of intervention
  Dose modifications (intensity or volume) in each session will be recorded. The number and percentage of dose modification will be calculated and provided.
Adverse Events | During 24 weeks of intervention
  Adverse events (safety and technical) in each session will be recorded. The number and percentage of each type of adverse event will be calculated and provided.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Irazusta, Prof, Principal Investigator — University of the Basque Country (UPV/EHU)
Locations (4):
- Spain (4):
  - Residencia Aspaldiko, Portugalete, Bizkaia
  - Residencia Nuestra Señora de Begoña, Santurtzi, Bizkaia
  - Residencia Albiz Santiago LLanos, Sestao, Bizkaia
  - Fundación Miranda, Barakaldo, Vizcaya

IPD SHARING:
Plan to Share IPD: Yes
The anonymized data may be shared, following a reasoned proposal
Supporting Information: Study Protocol
Access Criteria: The protocol data may be shared, following a reasoned proposal

REFERENCES:
- [Background] Llinas-Regla J, Vilalta-Franch J, Lopez-Pousa S, Calvo-Perxas L, Torrents Rodas D, Garre-Olmo J. The Trail Making Test. Assessment. 2017 Mar;24(2):183-196. doi: 10.1177/1073191115602552. Epub 2016 Jul 28. PMID 26318386
- [Background] Martínez de la Iglesia J, Onís-Vilches MC, Dueñas-Herrero R, et ál. Versión española del cuestionario de Yesavage abreviado (GDS) para el despistaje de depresión en mayores de 65 años: adaptación y validación. Medifam. 2002; 12(10):620.
- [Background] Rikli, R.E., Jones, C.J. Senior Fitness Test. Champaign: Human Kinetics; 2001. (ISBN 0-7360- 3356-3364).
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Wechsler D. WAIS III: escala de inteligencia de Wechsler para adultos-III manual técnico. Madrid: TEA; 1999
- [Background] Herdman M, Badia X, Berra S. [EuroQol-5D: a simple alternative for measuring health-related quality of life in primary care]. Aten Primaria. 2001 Oct 15;28(6):425-30. doi: 10.1016/s0212-6567(01)70406-4. No abstract available. Spanish. PMID 11602124
- [Background] Moreno, J. A., González-Cutre, D., Chillón, M., y Parra, N. (2008). Adaptación a la educación física de la escala de las necesidades psicológicas básicas en el ejercicio. Revista Mexicana de Psicología, 25(2), 295-303
- [Background] Hernández-Pozo, M., Macías, D., Calleja, N., Cerezo, S., & del Valle Chauvet, C. (2008). Propiedades psicometricas del inventario Zung del estado de ansiedad con mexicanos. Psychologia. Avances de la disciplina, 2(2), 19-46.
- [Background] Vazquez C, Duque A, Hervas G. Satisfaction with life scale in a representative sample of Spanish adults: validation and normative data. Span J Psychol. 2013;16:E82. doi: 10.1017/sjp.2013.82. PMID 24230945
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Pin TW. Psychometric properties of 2-minute walk test: a systematic review. Arch Phys Med Rehabil. 2014 Sep;95(9):1759-75. doi: 10.1016/j.apmr.2014.03.034. Epub 2014 May 9. PMID 24814460
- [Background] Fess EE. Grip strength. In: Casanova JS, editor. Clinical assessment recommendations, 2nd ed. Chicago: American Society of Hand Therapists; 1992. pp. 41-45.
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Kaehr E, Visvanathan R, Malmstrom TK, Morley JE. Frailty in nursing homes: the FRAIL-NH Scale. J Am Med Dir Assoc. 2015 Feb;16(2):87-9. doi: 10.1016/j.jamda.2014.12.002. Epub 2014 Dec 31. No abstract available. PMID 25556303
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Rodriguez-Larrad A, Arrieta H, Rezola C, Kortajarena M, Yanguas JJ, Iturburu M, Susana MG, Irazusta J. Effectiveness of a multicomponent exercise program in the attenuation of frailty in long-term nursing home residents: study protocol for a randomized clinical controlled trial. BMC Geriatr. 2017 Feb 23;17(1):60. doi: 10.1186/s12877-017-0453-0. PMID 28231827